CLINICAL TRIAL: NCT03265184
Title: Effects of Green Coffee Extract Supplementation on Oxidative Stress, Systemic and Vascular Inflammation in Patients With Metabolic Syndrome: A Randomized Clinical Trial
Brief Title: Green Coffee Extract Supplementation and Oxidative Stress, Systemic and Vascular Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, National Nutrition and Food Technology Research Institute, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NationalNFTI1355
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): 400 mg green coffee extract capsules twice per day for 8 weeks The Green coffee extract is standardised with 45% total chlorogenic acid by HPLC
  Interventions: Dietary Supplement: green coffee extract
- placebo group (Placebo Comparator): placebo capsules twice per day for 8 weeks have identical appearance to Green coffee extract capsules and contain starch
  Interventions: Dietary Supplement: green coffee extract

INTERVENTIONS:
Dietary Supplement: green coffee extract — Patients in treatment group take 400 mg GCE supplements twice a day for tow month

SUMMARY:
Metabolic syndrome (Mets) is defined as the collection of risk factors contributing to type 2 diabetes mellitus and cardiovascular disease. Mets is accompanied by oxidative stress and low-grade inflammation. Green coffee is rich in polyphenols called chlorogenic acids (CGA) which possess anti-inflammatory and anti-oxidative characteristics. Thus, we carried out this trial to examine green coffee extract (GCE) effects on oxidative stress, systemic and vascular inflammation in patients having Mets

ELIGIBILITY:
Inclusion Criteria:

* body mass index of over 25, waist circumference >102 cm in men or >88 cm in women,Fasting blood glucose >100 mg/dL, Triglycerides (TG) > 150 mg/dL, High density lipoprotein cholesterol (HDL-C) <50 in women or <40 in men, Systolic blood pressure (SBP) >130 mmHg and diastolic blood pressure (DBP) >85mmHg

Exclusion Criteria:

* insulin administration for diabetes control, having hypo- or hyperthyroidism, renal failure or other chronic diseases, regular coffee consumption, pregnancy, breastfeeding, taking estrogen, progesterone, corticosteroids, weight loss supplements and obeying unusual weight loss plans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
intercellular adhesion molecule-1 (ICAM-1) | 8 weeks
interleukin-6 (IL-6) | 8 weeks
high sensitivity C-reactive protein (hs-CRP) | 8 weeks
malondialdehyde (MDA) | 8 weeks